CLINICAL TRIAL: NCT04883957
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of Bcl-2 Inhibitor BGB-11417 in Adult Patients With Mature B-cell Malignancies
Brief Title: Study of BGB-11417 in Adult Participants With Mature B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-102; CTR20211017 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Mature B-cell Malignancies
Keywords: BGB-11417; Bcl-2; Pharmacokinetics; RP2D; MTD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: R/R NHL (Experimental): Participants with R/R NHL, including follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), marginal zone lymphoma (MZL), or transformed NHL, will receive oral BGB-11417 until the MTD (or maximum ascending dose [MAD]) and the RP2D can be determined.
  Interventions: Drug: BGB-11417
- Cohort B: R/R CLL/SLL (low tumor burden) (Experimental): Participants with low tumor burden R/R CLL/SLL will receive oral BGB-11417 until the MTD (or MAD) and the RP2D can be determined.
  Interventions: Drug: BGB-11417
- Cohort C: R/R CLL/SLL (high tumor burden) (Experimental): Participants in this cohort will not be enrolled until the RP2D for Cohort B is established. Participants will be treated with the monotherapy ramp-up schedule and the RP2D established in Cohort B.
  Interventions: Drug: BGB-11417

INTERVENTIONS:
Drug: BGB-11417 — Film-coated tablets administered orally as specified in the treatment arm.
  Other Names: Sonrotoclax

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of BGB-11417 monotherapy, define the maximum tolerated dose (MTD) or maximum administered dose and the recommended Phase 2 dose (RP2D) of BGB-11417 monotherapy for the selected B-cell malignancy dose finding cohorts, and evaluate the safety and tolerability of the ramp-up dosing schedule in the evaluated disease types.

DETAILED DESCRIPTION:
This study will have 3 cohorts for determining a monotherapy MTD and ramp-up schedule: Cohort A, participants with relapsed/refractory B-cell non-Hodgkin lymphoma (R/R NHL); Cohort B, participants with R/R chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) with low tumor burden; Cohort C, participants with R/R CLL/SLL with high tumor burden.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis of only one of the following:

   Cohort A

   a. Marginal Zone Lymphoma

   i. R/R extranodal, splenic or nodal disease defined as disease that has relapsed after, or been refractory to, ≥ 1 line of anti-CD20 antibody-based chemoimmunotherapy for ≥ 2 consecutive cycles, and no effective standard therapy for MZL is available per investigator's assessment.

   ii. Active disease requiring treatment.

   b. Follicular Lymphoma

   i. R/R FL (Grade 1, 2 or 3a based on the WHO 2008 classification of tumors of hematopoietic and lymphoid tissue) and defined as disease that has relapsed after, or been refractory to, ≥ 1 line of anti-CD20 antibody-based chemoimmunotherapy for ≥ 2 consecutive cycles, and no effective standard therapy for FL is available per investigator's assessment.

   ii. Active disease requiring treatment.

   c. Diffuse Large B-cell Lymphoma

   i. R/R DLBCL defined as disease that relapsed after, or been refractory to, at least one line of anti-CD20 antibody based chemoimmunotherapy for ≥ 2 consecutive cycles, and no effective standard therapy for DLBCL is available per investigator's assessment.

   ii. Active disease requiring treatment.

   d. Transformed indolent B-cell NHL

   i. Any lymphoma otherwise eligible for Cohort A that has transformed into a more aggressive lymphoma. Patients with transformation from CLL or SLL (Richter's transformation) are not eligible for Cohort A.

   ii. Active disease requiring treatment.

   Cohorts B and C

   a. CLL/SLL diagnosis that meets the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria:

   i. R/R disease defined as disease that has relapsed after, or been refractory to, ≥ 1 line of standard therapy for ≥ 2 consecutive cycles, and no effective standard therapy is available per investigator's assessment.

   ii. Requiring treatment based on IWCLL criteria.
2. Measurable disease by computed tomography/magnetic resonance imaging, defined as:

   1. CLL: At least 1 lymph node > 1.5 centimeters (cm) in longest diameter and measurable in 2 perpendicular dimensions. For Cohort B, participants should not meet with the definition of high tumor burden, which is required for participants enrolled in Cohort C.
   2. DLBCL, FL, MZL, SLL: At least 1 lymph node > 1.5 cm in longest diameter OR 1 extranodal lesion > 1.0 cm in the longest diameter, measurable in 2 perpendicular dimensions. For MZL isolated splenomegaly is considered to indicate measurable disease for this study. For SLL, participants in Cohort B should not meet with the definition of high tumor burden, which is required for participants enrolled in Cohort C.

Key Exclusion Criteria:

1. Prior malignancy (other than the disease under study) within the past 2 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score ≤ 6 prostate cancer.
2. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of safety or efficacy results.
3. Known central nervous system involvement by lymphoma/leukemia.
4. Known plasma cell neoplasm, prolymphocytic leukemia, history of or currently suspected Richter's syndrome.
5. Prior autologous stem cell transplant unless ≥ 3 months after transplant; or prior chimeric cell therapy unless ≥ 6 months after cell infusion.
6. Prior allogeneic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
MTD Of BGB-11417 As Recommended By The Bayesian Logistic Regression Model Or The MAD | Approximately 3 years
RP2D Of BGB-11417 | Approximately 3 years
  The RP2D will be decided by the sponsor and based on the safety monitoring committee recommendation considering totality of data.
Incidence And Severity Of Treatment-emergent Adverse Events, Serious Adverse Events, Adverse Events (AEs) Leading To Discontinuation, And Dose-Limiting Toxicities (DLTs) | Approximately 3 years
  All AEs, including DLT events, will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 (or the Grading Scale for Hematologic Toxicity in CLL Studies as appropriate).
Incidence And Severity Of Tumor Lysis Syndrome-relevant Events | Approximately 3 years

SECONDARY OUTCOMES:
Pharmacokinetics (PK) As Assessed By Maximum Observed Plasma Concentration (Cmax) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To The Time Of The Last Quantifiable Concentration (AUC0-t) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To Infinity (AUC0-inf) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Time To Maximum Observed Plasma Concentration (tmax) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Terminal Half-life (t1/2) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Apparent Total Clearance Of Drug From Plasma After Oral Administration (CL/F) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Apparent Volume Of Distribution (Vz/F) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Area Under The Plasma Concentration Time Curve From Time 0 To Last Measurable Concentration At Steady State (AUClast,ss) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Maximum Observed Plasma Concentration At Steady State (Cmax,ss) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Trough Concentration At Steady State (Ctrough,ss) Of BGB-11417 | Up to 24 hours postdose
PK As Assessed By Time To Maximum Observed Plasma Concentration At Steady State (tmax,ss) Of BGB-11417 | Up to 24 hours postdose
Overall Response Rate (ORR) Of BGB-11417 Monotherapy | Approximately 3 years
  ORR will be assessed per disease-specific response assessment guidelines as determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Zhang, M.D., Study Director — BeiGene (Suzhou) Co., Ltd.
Locations (11):
- China (11):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Peoples Hospital, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes